CLINICAL TRIAL: NCT04983173
Title: The Impact of the Intensity of Ovarian Stimulation on Embryo Quality in Predicted Suboptimal Responders. A Randomized Controlled Trial
Brief Title: INTEnsity of ovariaN Stimulation and Embryo Quality
Acronym: INTENS-EQ
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-IEQ-2021-03; 2021-000941-42 (EudraCT Number)
Record Dates: First submitted 2021-07-05; First posted 2021-07-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Clomiphene Citrate (CC) + rFSH (Experimental): Ovarian Stimulation with CC+rFSH
  Interventions: Drug: Ovarian Stimulation with CC+rFSH
- rFSH (Active Comparator): Ovarian Stimulation with rFSH
  Interventions: Drug: Ovarian Stimulation with rFSH

INTERVENTIONS:
Drug: Ovarian Stimulation with CC+rFSH — : CC 50 mg/day (Omifin®) + rFSH 150 IU (Ovaleap®) GnRH antagonist: ganirelix 0.25 mg (Orgalutran®) Recombinant human chorionic gonadotropin (rhCG) 250 μg (Ovitrelle®) micronized progesterone 200 mg 3id (Utrogestan®)
  Arms: Experimental: Clomiphene Citrate (CC) + rFSH
Drug: Ovarian Stimulation with rFSH — rFSH 300 IU rFSH (Ovaleap®) GnRH antagonist: ganirelix 0.25 mg (Orgalutran®) Recombinant human chorionic gonadotropin (rhCG) 250 μg (Ovitrelle®) micronized progesterone 200 mg 3id (Utrogestan®)
  Arms: rFSH

SUMMARY:
The management of suboptimal ovarian responders remains a challenging task in IVF. These patients are frequently managed with an intense stimulation protocol of ovarian stimulation in order obtain the maximum number of embryos and, therefore, maximize the cumulative live birth rate. However, the concept of "the more the better" has been recently defied by the one of "mild stimulation". Defenders of this protocol state that with mild stimulation only the best quality oocytes are allowed to grow and, therefore, higher quality embryos will be obtained. However, the impact of the intensity of ovarian stimulation on embryo quality is far from consensual. Moreover, its effect on early embryo development has never been evaluated.

Therefore, the investigators set out to perform this randomized controlled trial comparing the number of GQB and the morphokinetic parameters of early embryo development in infertile patients undergoing two different intensities of ovarian stimulation, a milder approach (CC plus 150 IU daily dose of rFSH) and a more intense approach (300 IU daily dose of rFSH).

DETAILED DESCRIPTION:
Despite the lack of a consistent definition for "mild stimulation" (MS), the International Society for Mild Approaches in Assisted Reproduction defined it as a protocol performed with gonadotropins, alone or with oral compounds, at lower doses or for a shorter duration, with the aim of achieving 2-7 oocytes. One of the strategies proposed for MS is the use of Clomiphene Citrate (CC). CC acts as a selective estrogen-receptor modulator. By blocking estrogen receptors in the hypothalamic arcuate nucleus, it increases the production of gonadotropin-releasing hormone (GnRH) and, as a result, FSH and luteinizing hormone (LH). Moreover, CC increases the pituitary sensitivity to GnRH and granulosa cell sensitivity to pituitary gonadotropins. Taking these actions into account, several protocols have adopted a combination of CC and exogenous gonadotropins with the aim of improving follicular recruitment and, therefore, ovarian response to stimulation, in patients undergoing in vitro fertilization (IVF). The available evidence has allowed for the inclusion of CC in international guidelines as a treatment option, alone or in combination with gonadotropins, equally recommended in the management of poor responders when compared to gonadotropin stimulation alone.

The concept behind MS is that, with this approach, only the healthier follicles with higher quality oocytes are allowed to grow. Proponents of this protocol state that MS reduces the risk of multiple pregnancy and ovarian hyperstimulation syndrome (OHSS), as well as patient dropout rate and treatment costs. However, evidence regarding clinical outcomes is far from consensual. The best available evidence regarding MS in predicted poor responders comes from the OPTIMIST trial, showing no difference in the cumulative live birth rates when a mild approach, using 150 IU of rFSH, was compared to an individualized protocol of 225/450 IU rFSH. However, several methodological inconsistencies have been pointed out in this randomized controlled trial. In particular, a black hole was left in the management of predicted low responders with an intermediate prognosis (antral follicle count between 8-10), taking into account the allowance for dose adjustments in the second cycle in the 150 IU group. Considering that the control group was treated with rFSH 225 IU daily, a comparison of two identical doses might have been provided.

Evidence regarding the effect of MS on embryo quality is also conflicting. Baart et al. first reported a lower aneuploidy rate following MS when compared to conventional protocols and concluded that mitotic segregation errors might increase with growing gonadotropin dosages. However, this has not been confirmed in recent studies. As for the number of good quality embryos, while previous studies have shown no difference regarding MS and conventional protocols, Vermey et al found a positive correlation between the number of retrieved oocytes and the embryo quality.

Although these previous studies provide some valuable information, the heterogeneity of the available evidence cannot be disregarded. Moreover, to the best our knowledge, the effect of the intensity of ovarian stimulation on early embryo development has not been previously described. Therefore, the investigators set out to perform this randomized controlled trial comparing the number of good quality blastocysts (GQB) and morphokinetic parameters of early embryo development in patients with a predicted suboptimal ovarian response undergoing two different intensities of ovarian stimulation, a milder (CC 50 mg/day from cycle D2-6 + rFSH 150 IU daily from D2 onwards) and a more intense approach (300 IU daily dose of rFSH starting on cycle D2).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign the Patient Consent Form and adhere to study visitation schedule
* Antral follicle count (AFC) ≥ 5 and ≤ 10
* Anti-Mullerian hormone (AMH) ≤1.5 ng/ml (AMH result of up to one year will be valid)
* Age ≥ 35 years and ≤40 years
* BMI ≥18.5 and <25 kg/m2

Exclusion Criteria:

* AFC >10
* History of untreated autoimmune, endocrine or metabolic disorders
* Contraindication for hormonal treatment
* Preimplantation genetic diagnosis cycles
* Severe male factor (sperm concentration <5 M/mL)
* Recent history of severe disease requiring regular treatment (clinically significant concurrent medical condition that could compromise subject safety or interfered with the trial assessment and patients with any contraindication of being pregnant).

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of good quality blastocysts | Until 5, 6 or 7 days after oocyte pick-up

SECONDARY OUTCOMES:
Change in Progesterone values | days 1, 6, 8, 10 and the day of ovulation triggering
Change in Estradiol values | days 1, 6, 8, 10 and the day of ovulation triggering
Change in FSH Values | days 1, 6, 8, 10 and the day of ovulation triggering
Change in LH values | days 1, 6, 8, 10 and the day of ovulation triggering
Length of ovarian stimulation | 7 -20 days from initiation of ovarian stimulation
Number of oocytes retrieved | 7 -20 days from initiation of ovarian stimulation
Number of mature oocytes (MIIs) retrieved | 7 -20 days from initiation of ovarian stimulation
Follicle to Oocyte Index (FOI) | 7 -20 days from initiation of ovarian stimulation
  ratio of the number of preovulatory follicles and the number of antral follicles available at the start of stimulation
Total dose of rFSH | 7 -20 days from initiation of ovarian stimulation
Follicular Output Rate (FORT) | 7 -20 days from initiation of ovarian stimulation
  ratio of the number of preovulatory follicles and the number of antral follicles available at the start of stimulation
Cycle cancelation rate | Until 15 days after the beginning of ovarian stimulation
  when no follicle has adequate maturation, or the follicle is lost due to spontaneous LH surge
Reason for cycle cancelation | Until 15 days after the beginning of ovarian stimulation
Fertilization rate | One day after oocyte pick-up
Time of appearance of the 2nd polar body (tPB2) | One day after oocyte pick-up
Time of pronuclei appearance (tPNa) | One day after oocyte pick-up
Evaluation of both pronuclei (PN) | One day after oocyte pick-up
Time of pronuclei disappearance (tPNf) | Day 2 after insemination
Time of division from 2 to 8 cells (t2, t3, t4, t5, t6, t7, t8) | Until Day 2 Day 3 after insemination
Time of compactation (tSC) | Until Day 3 Day 6 after insemination
Time of morula (tM) | Until Day 3 Day 6 after insemination
Time of cavitation (tSB) | Until 5, 6 or 7 days after insemination
Time of full blastulation (tB) | Until 5, 6 or 7 days after insemination
Time of expanded blastocyst (tEB) | Until 5, 6 or 7 days after insemination
Time of hatched blastocyst (tHB) | Until 5, 6 or 7 days after insemination
Time of embryo discarding (tDead) | Until 7 days after insemination
Total number of embryos | Until 5, 6 or 7 days after insemination
Blastocyst formation rate | Until 5, 6 or 7 days after insemination
Number of embryos cryopreserved | Until 5, 6 or 7 days after insemination
Embryo stage (D5, D6, D7) | Until 5, 6 or 7 days after insemination
Clinical pregnancy rate | 5 to 6 weeks after oocyte pick-up
  defined as a viable intrauterine pregnancy of at least 8-10 weeks duration confirmed on an ultrasound scan
Ongoing pregnancy rate | 8 to 10 weeks after oocyte pick-up

OTHER OUTCOMES:
Ovarian hyperstimulation syndrome (OHSS) (percent) | Until 15 days after the end of ovarian stimulation
  Number of subjects with OHSS during the ovarian stimulation period and their severity
Miscarriages | before completion of 12 weeks of gestation
  any spontaneous abortion that occurred after confirmation of clinical pregnancy
Incidence of adverse events and serious adverse events | Until 15 days after the end of ovarian stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD PhD, Study Chair — Hospital Universitari Dexeus; Ana Neves, MD, Principal Investigator — Hospital Universitari Dexeus
Locations (1):
- Salud de la Mujer Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nargund G, Fauser BC, Macklon NS, Ombelet W, Nygren K, Frydman R; Rotterdam ISMAAR Consensus Group on Terminology for Ovarian Stimulation for IVF. The ISMAAR proposal on terminology for ovarian stimulation for IVF. Hum Reprod. 2007 Nov;22(11):2801-4. doi: 10.1093/humrep/dem285. Epub 2007 Sep 12. PMID 17855409
- [Background] Dickey RP, Holtkamp DE. Development, pharmacology and clinical experience with clomiphene citrate. Hum Reprod Update. 1996 Nov-Dec;2(6):483-506. doi: 10.1093/humupd/2.6.483. PMID 9111183
- [Background] Bechtejew TN, Nadai MN, Nastri CO, Martins WP. Clomiphene citrate and letrozole to reduce follicle-stimulating hormone consumption during ovarian stimulation: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2017 Sep;50(3):315-323. doi: 10.1002/uog.17442. Epub 2017 Aug 10. PMID 28236310
- [Background] Kamath MS, Maheshwari A, Bhattacharya S, Lor KY, Gibreel A. Oral medications including clomiphene citrate or aromatase inhibitors with gonadotropins for controlled ovarian stimulation in women undergoing in vitro fertilisation. Cochrane Database Syst Rev. 2017 Nov 2;11(11):CD008528. doi: 10.1002/14651858.CD008528.pub3. PMID 29096046
- [Background] ESHRE Reproductive endocrinology guidelines group. Ovarian Stimulation for IVF / ICSI - Guideline of the European Society of Human Reproduction and Embryology. Belgium: ESHRE; 2019
- [Background] Zhang JJ, Merhi Z, Yang M, Bodri D, Chavez-Badiola A, Repping S, van Wely M. Minimal stimulation IVF vs conventional IVF: a randomized controlled trial. Am J Obstet Gynecol. 2016 Jan;214(1):96.e1-8. doi: 10.1016/j.ajog.2015.08.009. Epub 2015 Aug 8. PMID 26259908
- [Background] Verberg MF, Eijkemans MJ, Heijnen EM, Broekmans FJ, de Klerk C, Fauser BC, Macklon NS. Why do couples drop-out from IVF treatment? A prospective cohort study. Hum Reprod. 2008 Sep;23(9):2050-5. doi: 10.1093/humrep/den219. Epub 2008 Jun 10. PMID 18544578
- [Background] Heijnen EM, Eijkemans MJ, De Klerk C, Polinder S, Beckers NG, Klinkert ER, Broekmans FJ, Passchier J, Te Velde ER, Macklon NS, Fauser BC. A mild treatment strategy for in-vitro fertilisation: a randomised non-inferiority trial. Lancet. 2007 Mar 3;369(9563):743-749. doi: 10.1016/S0140-6736(07)60360-2. PMID 17336650
- [Background] Aleyamma TK, Kamath MS, Muthukumar K, Mangalaraj AM, George K. Affordable ART: a different perspective. Hum Reprod. 2011 Dec;26(12):3312-8. doi: 10.1093/humrep/der323. Epub 2011 Oct 10. PMID 21987524
- [Background] Paulson RJ, Fauser BCJM, Vuong LTN, Doody K. Can we modify assisted reproductive technology practice to broaden reproductive care access? Fertil Steril. 2016 May;105(5):1138-1143. doi: 10.1016/j.fertnstert.2016.03.013. Epub 2016 Apr 4. PMID 27054309
- [Background] Polyzos NP, Popovic-Todorovic B. SAY NO to mild ovarian stimulation for all poor responders: it is time to realize that not all poor responders are the same. Hum Reprod. 2020 Sep 1;35(9):1964-1971. doi: 10.1093/humrep/deaa183. PMID 32830232
- [Background] van Tilborg TC, Torrance HL, Oudshoorn SC, Eijkemans MJC, Koks CAM, Verhoeve HR, Nap AW, Scheffer GJ, Manger AP, Schoot BC, Sluijmer AV, Verhoeff A, Groen H, Laven JSE, Mol BWJ, Broekmans FJM; OPTIMIST study group. Individualized versus standard FSH dosing in women starting IVF/ICSI: an RCT. Part 1: The predicted poor responder. Hum Reprod. 2017 Dec 1;32(12):2496-2505. doi: 10.1093/humrep/dex318. PMID 29121326
- [Background] Verberg MF, Eijkemans MJ, Macklon NS, Heijnen EM, Baart EB, Hohmann FP, Fauser BC, Broekmans FJ. The clinical significance of the retrieval of a low number of oocytes following mild ovarian stimulation for IVF: a meta-analysis. Hum Reprod Update. 2009 Jan-Feb;15(1):5-12. doi: 10.1093/humupd/dmn053. PMID 19091754
- [Background] Matsaseng T, Kruger T, Steyn W. Mild ovarian stimulation for in vitro fertilization: are we ready to change? A meta-analysis. Gynecol Obstet Invest. 2013;76(4):233-40. doi: 10.1159/000355980. Epub 2013 Nov 2. PMID 24192422
- [Background] Sterrenburg MD, Veltman-Verhulst SM, Eijkemans MJ, Hughes EG, Macklon NS, Broekmans FJ, Fauser BC. Clinical outcomes in relation to the daily dose of recombinant follicle-stimulating hormone for ovarian stimulation in in vitro fertilization in presumed normal responders younger than 39 years: a meta-analysis. Hum Reprod Update. 2011 Mar-Apr;17(2):184-96. doi: 10.1093/humupd/dmq041. Epub 2010 Sep 15. PMID 20843965
- [Background] Baart EB, Martini E, Eijkemans MJ, Van Opstal D, Beckers NG, Verhoeff A, Macklon NS, Fauser BC. Milder ovarian stimulation for in-vitro fertilization reduces aneuploidy in the human preimplantation embryo: a randomized controlled trial. Hum Reprod. 2007 Apr;22(4):980-8. doi: 10.1093/humrep/del484. Epub 2007 Jan 4. PMID 17204525
- [Background] La Marca A, Minasi MG, Sighinolfi G, Greco P, Argento C, Grisendi V, Fiorentino F, Greco E. Female age, serum antimullerian hormone level, and number of oocytes affect the rate and number of euploid blastocysts in in vitro fertilization/intracytoplasmic sperm injection cycles. Fertil Steril. 2017 Nov;108(5):777-783.e2. doi: 10.1016/j.fertnstert.2017.08.029. Epub 2017 Oct 4. PMID 28987789
- [Background] Wu Q, Li H, Zhu Y, Jiang W, Lu J, Wei D, Yan J, Chen ZJ. Dosage of exogenous gonadotropins is not associated with blastocyst aneuploidy or live-birth rates in PGS cycles in Chinese women. Hum Reprod. 2018 Oct 1;33(10):1875-1882. doi: 10.1093/humrep/dey270. PMID 30137360
- [Background] Venetis CA, Tilia L, Panlilio E, Kan A. Is more better? A higher oocyte yield is independently associated with more day-3 euploid embryos after ICSI. Hum Reprod. 2019 Jan 1;34(1):79-83. doi: 10.1093/humrep/dey342. PMID 30476100
- [Background] Irani M, Canon C, Robles A, Maddy B, Gunnala V, Qin X, Zhang C, Xu K, Rosenwaks Z. No effect of ovarian stimulation and oocyte yield on euploidy and live birth rates: an analysis of 12 298 trophectoderm biopsies. Hum Reprod. 2020 May 1;35(5):1082-1089. doi: 10.1093/humrep/deaa028. PMID 32348476
- [Background] Ghosh Dastidar S, Maity S, Ghosh Dastidar B. Reappraisal of IVF stimulation in good prognosis patients - a prospective randomized study to compare mild versus standard long protocol. Fertil Steril [Internet]. 2010;94(4):S28. Available from: http://dx.doi.org/10.1016/j.fertnstert.2010.07.108
- [Background] Golan A, Weissman A. Symposium: Update on prediction and management of OHSS. A modern classification of OHSS. Reprod Biomed Online. 2009 Jul;19(1):28-32. doi: 10.1016/s1472-6483(10)60042-9. PMID 19573287
- [Background] Hohmann FP, Macklon NS, Fauser BC. A randomized comparison of two ovarian stimulation protocols with gonadotropin-releasing hormone (GnRH) antagonist cotreatment for in vitro fertilization commencing recombinant follicle-stimulating hormone on cycle day 2 or 5 with the standard long GnRH agonist protocol. J Clin Endocrinol Metab. 2003 Jan;88(1):166-73. doi: 10.1210/jc.2002-020788. PMID 12519847
- [Background] Datta AK, Maheshwari A, Felix N, Campbell S, Nargund G. Mild versus conventional ovarian stimulation for IVF in poor, normal and hyper-responders: a systematic review and meta-analysis. Hum Reprod Update. 2021 Feb 19;27(2):229-253. doi: 10.1093/humupd/dmaa035. PMID 33146690
- [Background] Vermey BG, Chua SJ, Zafarmand MH, Wang R, Longobardi S, Cottell E, Beckers F, Mol BW, Venetis CA, D'Hooghe T. Is there an association between oocyte number and embryo quality? A systematic review and meta-analysis. Reprod Biomed Online. 2019 Nov;39(5):751-763. doi: 10.1016/j.rbmo.2019.06.013. Epub 2019 Jul 3. PMID 31540848
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182
- [Background] ESHRE Special Interest Group of Embryology and Alpha Scientists in Reproductive Medicine. Electronic address: coticchio.biogenesi@grupposandonato.it. The Vienna consensus: report of an expert meeting on the development of ART laboratory performance indicators. Reprod Biomed Online. 2017 Nov;35(5):494-510. doi: 10.1016/j.rbmo.2017.06.015. Epub 2017 Aug 4. PMID 28784335
- [Background] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Fertil Steril. 2017 Sep;108(3):393-406. doi: 10.1016/j.fertnstert.2017.06.005. Epub 2017 Jul 29. PMID 28760517
- [Background] Montoya-Botero P, Martinez F, Rodriguez-Purata J, Rodriguez I, Coroleu B, Polyzos NP. Erratum. The effect of type of oral contraceptive pill and duration of use on fresh and cumulative live birth rates in IVF/ICSI cycles. Hum Reprod. 2021 Mar 18;36(4):1159-1161. doi: 10.1093/humrep/deaa358. No abstract available. PMID 33515004
- See also: Department of Obstetrics, Gynaecology and Reproduction Hospital Universitari Quiron Dexeus — http://www.dexeus.com